CLINICAL TRIAL: NCT05898217
Title: Relative Absorption of Fat-soluble Vitamin D and Minerals From Select Plant-based Milks in Human Subjects
Brief Title: Vitamin and Mineral Absorption From Milk and PBMAs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2023-83
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Nutrition; Healthy
Keywords: calcium; vitamin D; potassium; magnesium; dairy; plant-based
MeSH Terms: interventions — Milk; Soy Milk

STUDY DESIGN:
Intervention Model Description: 4 groups, each are assigned to one week of drinking fluid milk, almond milk, soy milk, or oat milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dairy Milk (Active Comparator): Participants will drink 16 oz of dairy milk daily for the duration of the study.
  Interventions: Other: Dairy Milk
- Soy Milk (Active Comparator): Participants will drink 16 oz of soy milk daily for the duration of the study.
  Interventions: Other: Soy Milk
- Almond Milk (Active Comparator): Participants will drink 16 oz of almond milk daily for the duration of the study.
  Interventions: Other: Almond Milk
- Oat Milk (Active Comparator): Participants will drink 16 oz of oat milk daily for the duration of the study.
  Interventions: Other: Oat Milk

INTERVENTIONS:
Other: Dairy Milk — Daily, each participant will consume 16 oz of the type of milk (plant based or dairy) two which they are randomized.
  Arms: Dairy Milk
Other: Soy Milk — Daily, each participant will consume 16 oz of the type of milk (plant based or dairy) two which they are randomized.
  Arms: Soy Milk
Other: Almond Milk — Daily, each participant will consume 16 oz of the type of milk (plant based or dairy) two which they are randomized.
  Arms: Almond Milk
Other: Oat Milk — Daily, each participant will consume 16 oz of the type of milk (plant based or dairy) two which they are randomized.
  Arms: Oat Milk

SUMMARY:
Plant-based milk alternatives (PBMAs) are a popular alternative to cow's milk. The different types of PBMAs on the market shelf include almond, oat, soy, coconut, cashew, pea, hemp, and rice. Among these, PBMA made from almonds, oats and soy are the most popular in North America. Though PBMAs are designed to mimic cow's milk in terms of color, they often have a very different nutrition profile. In order to better substitute for cow's milk, PBMAs often have added vitamins and minerals, as well as added sugars and flavorings to improve flavor.

This study will test how well certain nutrients (vitamin D, calcium, potassium, and magnesium) are absorbed by the body after intake of milk and PBMAs. Nutrient absorption will be measured using blood samples after short term intake (from 1 hours to 1 week) of almond, soy, and oat milk, and compare it to cow's milk. Participants in the study will avoid all fluid dairy products and vitamin-D supplemented foods for three weeks and then be asked to consume either almond, soy, oat, or cow's milk for one week.

All participants will visit the Clinical Nutrition Research Center (CNRC) four times over the course of about one month. These visits include a screening and pre-study visit (1.5 hrs), a pick-up visit (30 min), one long study day visit (~11 hours), and two shorter follow up study day visits (1 hr).

DETAILED DESCRIPTION:
The study has several objectives:

1. The main objective is to conduct a short-term research trial to understand the relative absorption of key micronutrients (Vitamin D, calcium, potassium and magnesium) from select PBMAs.
2. Develop and validate a method for measuring the amount of Vitamin D in blood.
3. Develop and validate a method for measuring the amount of magnesium, calcium, and potassium in blood and in urine.
4. Compare the amount of vitamin D and minerals in blood of people assigned to drink cow's milk to people who those assigned to drink plant-based milk alternatives.

This study will test how well certain nutrients (Vitamin D, calcium, potassium, and magnesium) are absorbed by the body after intake. We will examine nutrient absorption after short term intake (from 1 hour to 1 week) of almond, soy, and oat milk, and compare it to cow's milk. Participants in the study will avoid all fluid dairy products and any dairy or foods fortified with vitamin D for three weeks and then will be asked to consume either almond, soy, oat, or cow's milk for one week. All participants will visit the Clinical Nutrition Research Center (CNRC) at least five times over the course of about one month. The visits will proceed as follows:

1. Participants will come to IIT Mies campus for a screening visit. Blood pressure, blood sugar via finger prick, and anthropometric measurements (height, weight, body composition) will be taken. Women under age 60 will be asked for urine sample for pregnancy test. Participants who qualify will stay an additional 30 minutes for a prestudy visit where they will learn how to participate in the trial and schedule their study visits.
2. Standardized dinner pick up visit - participants will come to the IIT Mies campus to pick up a standardized dinner meal to eat before their Study Day 1 visit.
3. Study Day 1 Visit - Participants will have a catheter placed and a baseline blood draw will be performed. Participants will be randomized to one of four groups (almond milk, soy milk, oat milk, or cow's milk) and will drink 480 mL (16 oz) of that beverage. After the drink, blood will be collected via the catheter after 1 hour, 2 hours and then every 2 hours until hour 10. After 6 hours, participants will be given a light meal to alleviate hunger before the catheter is removed. Every hour, participants will be provided with 150 mL of distilled water to drink and urine will be collected after each blood draw. In total 50 mL of blood will be taken over the course of the day. After completing the study day, participants will be provided with a week's supply of the PBMA or milk and will be asked to drink 8 oz of the beverage 2x per day over the course of the following week while avoiding other dairy products.
4. Study Day 2 Visit: Participants will return to the IIT Mies campus 24 hours after the start of their Visit 1 and after a 10-12 hour fast. Anthropometric measurements, blood pressure, and blood sugar will be taken again. Then, 6 mL of blood will be drawn and urine collection will be performed.
5. Study Day 3 Visit: One week after Study Day Visit 1, participants will return to IIT Mies Campus. Anthropometric measurements, blood pressure, and blood sugar will be taken. Then, a fasting blood draw and urine collection will be performed. After fasting blood draw, participants will be given a snack. Total blood drawn will be 6 mL.

The blood and urine samples will be analyzed for specific nutrients and compared between the four randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 20.0-40.0 kg/m2, inclusive and a weight ≥ 110 lb. at the screening visit.
* Nonsmokers (Past smokers can be allowed if they have abstinence for minimum of 12 months)
* Judged to be in good health on the basis of the medical history i.e., no clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. proton pump inhibitors, anti-inflammatory drugs, antibiotics, vitamin D
* Willing to discontinue any multivitamin, vitamin or mineral supplements for three weeks immediately after date of the screening
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, records of food diary and GI tract questionnaire, sample collection procedures and study visit schedule)
* Able to maintain usual physical activity pattern
* Able to avoid vigorous physical activity, caffeine, and alcohol for 24 hours prior to and during study visit

Exclusion Criteria:

* Men and women who smoke or vape (including marijuana)
* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Men and women who have blood pressure >160 mmHg (systolic)/100 mmHg (diastolic) at screening visit
* Men and women who have fasting blood glucose concentration >125 mg/dL at screening visit
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
* Men and women with history of weight loss surgery or intestinal surgery which can impact digestion
* Men and women with osteoporosis
* Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g.,multivitamin, B complex supplement. Subjects may choose to go off dietary supplements (requires three week washout for multivitamin, three months for vitamin D supplements) before beginning the study.
* Men and women who have participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
* Men and women who have regularly taken Vitamin D supplements in the past 3 months
* Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
* Vegan or other extreme dietary regimens (e.g., Atkins diet, etc.) as judged by the investigator.
* Has a known intolerance or sensitivity to any ingredients in the study products
* Has used antibiotics within the previous 2 months
* Had colonoscopy within 3 months
* Has used prebiotics, probiotics, or drugs active on gastrointestinal motility, or a laxative of any class within 1 month
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d)
* Donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours i.e., working overnight (e.g. 3rd shift

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of vitamin D in plasma/serum | Collect data from 1 hour to 1 week post-consumption
  Measure the concentration of blood vitamin D postprandial and after short term (1 week) intake and compare between all arms.
Concentration of calcium, potassium, and magnesium in human serum and urine | Collect data from 1 hour to 1 week post-consumption
  Measure the concentration of blood and urine calcium, potassium, and magnesium postprandial and after short term (1 week) intake and compare between all arms.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Preiss, Study Director — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center Illinois Institute of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No